CLINICAL TRIAL: NCT03573778
Title: iHEAL in Context: Effectiveness of a Health Promotion Intervention for Women Who Have Experienced Intimate Partner Violence (iHEAL Trial)
Brief Title: IHEAL Trial: Effectiveness of a Health Promotion Intervention for Women Who Have Experienced Intimate Partner Violence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Collaborators: University of British Columbia (Other); University of New Brunswick (Other); McMaster University (Other); Johns Hopkins University (Other); Université de Montréal (Other); Public Health Agency of Canada (PHAC) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 111191
Record Dates: First submitted 2018-06-20; First posted 2018-06-29 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Intimate Partner Violence
Keywords: health; quality of life; safety; health promotion; intimate partner violence; domestic violence; confidence; control; nursing intervention

STUDY DESIGN:
Intervention Model Description: Randomized Controlled trial comparing active treatment to usual care
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iHEAL (Experimental): 10-18 visits (over 6 months) with a Registered Nurse
  Interventions: Behavioral: iHEAL
- Usual Care (Active Comparator): Information about Community Services
  Interventions: Behavioral: Information about Community Services

INTERVENTIONS:
Behavioral: iHEAL — Women work with a Registered Nurse in 10-18 visits (over 6 months) that focus on 6 inter-related 6 components (areas): Safeguarding, Managing Symptoms, Getting Basics, Cautiously Connecting, Regenerating Family, Renewing Self. Using a standard 3 phase process, and guided by 5 principles, the nurse discusses each of these components with the woman in order to identify the woman's needs, experiences and priorities. The nurse then provides personalized support to assist the woman in address the concerns that she sees as most important for her health and well-being; this support includes linking women to existing services if she chooses.
  Arms: iHEAL
Behavioral: Information about Community Services — Women are provided with information about community services appropriate for women experiencing intimate partner violence and consistent with what service providers might recommend (usual care). Women are encouraged to use this information as they see fit.
  Arms: Usual Care

SUMMARY:
Living with an abusive partner has many negative impacts on women's health, safety and the quality of their lives. These issues often continue when women separate, or take steps to separate, from an abusive partner, and can make it more difficult to create a new life. However, few supports are available to help women manage their health and other challenges around the time of separation.

The Intervention for Health Enhancement and Living (iHEAL) was specifically developed to support women at this time. In iHEAL, women work with a Registered Nurse on issues that affect that their health and well-being in 10 and 18 visits that take place in a safe, private location over a 6 month period. The woman decides which issues she would like to work on, with nurses providing personalized help and support that fits with the woman's needs, goals and wishes. This includes helping her connect to local services if she chooses.

The purpose of this study is to learn whether iHEAL can improve the health and quality of life of women who have separated, or are taking steps to separate, from an abusive partner. To do this, 280 Canadian women from 3 provinces will be offered either iHEAL nurse visits or information about community services that they can use on their own. All participants will complete online surveys when they first start the study and 6 12, and 18 months later to examine whether there are changes in their health, quality of life, confidence and/or control. We also want to learn whether iHEAL is more helpful for some groups of women and whether any benefits to women that are identified outweigh the costs of providing the intervention. A small group of ~30-40 women will be asked to take part in an interview about what is was like to take part in this study when they complete the trial so that we can learn how to further improve iHEAL.

DETAILED DESCRIPTION:
For a detailed description of the study rationale, hypotheses, research questions and methods, please see:

Ford-Gilboe, M., Varcoe, C., Scott-Storey, K. et al. Longitudinal effectiveness of a woman-led, nurse delivered health promotion intervention for women who have experienced intimate partner violence: iHEAL randomized controlled trial. BMC Public Health 24, 398 (2024). https://doi.org/10.1186/s12889-023-17578-4.

ELIGIBILITY:
Inclusion Criteria:

* Woman
* 19 years of age or older
* Able to speak, read and understand English
* Residing in specific communities in Ontario, British Columbia or New Brunswick
* Planning to remain in area for next 6 months
* Experienced physical, sexual, and/or psychological abuse, including coercive control from a current or former partner in the previous 12 months
* Planning to separate OR in the process of separating OR separated from an abusive partner in the previous 3 years
* Has access to the internet, and a safe computer, tablet, or smart phone
* Has a safe email address

Exclusion Criteria:

* Man
* Under 19 years of age
* Cannot read, speak, understand English
* Living outside of the selected study sites, or living in the area but planning to relocate within 6 months
* No experience of physical, sexual, or psychological abuse, including coercive control, from a current or former partner in the previous 12 months
* Planning to stay with an abusive partner OR separated more than 3 years ago
* No access to the internet, or safe computer, tablet or smart phone
* No access to safe email and mailing address

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Identifies as a woman
Enrollment: 331 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2020-04-24 (Actual); Study Completion 2021-05-22 (Actual)

PRIMARY OUTCOMES:
Changes in Quality of Life on the Quality of Life Scale (Sullivan) | baseline, 6 months
  9 item self-report measure developed to assess quality of life across domains important to women who have experienced intimate partner violence. Total scores range from 9 to 63. Higher scores reflect higher levels of quality of life.
Changes in PTSD Symptomology on the PTSD Checklist (Civilian Version) | baseline, 6 months
  17 item self-report measure of PTSD symptoms designed for use in community samples and to assess probability of meeting diagnostic criteria for PTSD.

SECONDARY OUTCOMES:
Changes in Quality of Life on the Quality of Life Scale (Sullivan) | baseline, 12 months
  9 item self-report measure developed to assess quality of life across domains important to women who have experienced intimate partner violence
Changes in Quality of Life on the Quality of Life Scale (Sullivan) | Baseline, 18 months
  9 item self-report measure developed to assess quality of life across domains important to women who have experienced intimate partner violence
Changes in PTSD Symptomology on the PTSD Checklist (Civilian Version) | Baseline, 12 months
  17 item self-report measure of PTSD symptoms designed for use in community samples and to assess probability of meeting diagnostic criteria for PTSD
Changes in PTSD Symptomology on the PTSD Checklist (Civilian Version) | Baseline, 18 months
  17 item self-report measure of PTSD symptoms designed for use in community samples and to assess probability of meeting diagnostic criteria for PTSD
Changes in Depressive Symptoms on the Center for Epidemiologic Studies Depression Scale, Revised (CESD-R). | Baseline, 6 months
  20 item self-report measure of depressive symptoms in community samples, including probability of meeting criteria for major depressive disorder. Total scores range from 0 to 60. Higher scores reflect higher levels of depressive symptoms.
Changes in Depressive Symptoms on the Center for Epidemiologic Studies Depression Scale, Revised | Baseline, 12 months
  20 item self-report measure of depressive symptoms in community samples, including probability of meeting criteria for major depressive disorder
Changes in Depressive Symptoms on the Center for Epidemiologic Studies Depression Scale, Revised | Baseline, 18 months
  20 item self-report measure of depressive symptoms in community samples, including probability of meeting criteria for major depressive disorder
Changes in Chronic Pain Disability on the Chronic Pain Grade (van Korff) | Baseline, 6 months
  7 item self-report measure of chronic pain intensity and disability, including 4 "grades" that capture level of disability (from no to high)
Changes in Chronic Pain Disability on the Chronic Pain Grade (van Korff) | Baseline, 12 months
  7 item self-report measure of chronic pain intensity and disability, including 4 "grades" that capture level of disability (from no to high)
Changes in Chronic Pain Disability on the Chronic Pain Grade (van Korff) | Baseline, 18 months
  7 item self-report measure of chronic pain intensity and disability, including 4 "grades" that capture level of disability (from no to high)
Changes in Personal Control on the Personal Agency Scale (Smith) | Baseline, 6 months
  8 item self-report scale that measures an individual's sense of control and efforts to act on their own behalf. Total scores range from 8 to 32. Higher scores reflect higher levels of personal agency.
Changes in Personal Control on the Personal Agency Scale (Smith) | Baseline, 12 months
  8 item self-report scale that measures an individual's sense of control and efforts to act on their own behalf. Total scores range from 8 to 32. Higher scores reflect higher levels of personal agency.
Changes in Personal Control on the Personal Agency Scale (Smith) | Baseline, 18 months
  8 item self-report scale that measures an individual's sense of control and efforts to act on their own behalf. Total scores range from 8 to 32. Higher scores reflect higher levels of personal agency.
Changes in Confidence (self-efficacy) on investigator-developed scale | Baseline, 6 months
  10 item self-report scale that measures women's confidence in engaging in a set of actions that fit with key goals of the iHEAL on 100 mm visual analogue scales. total scores range from 0 to 100. Higher scores reflect higher levels of confidence.
Changes in Confidence (self-efficacy) on investigator-developed scale | Baseline, 12 months
  10 item self-report scale that measures women's confidence in engaging in a set of actions that fit with key goals of the iHEAL on 100 mm visual analogue scales. Total scores range from 0 to 100. Higher scores reflected higher levels of confidence.
Changes in Confidence (self-efficacy) on investigator-developed scale | Baseline, 18 months
  10 item self-report scale that measures women's confidence in engaging in a set of actions that fit with key goals of the iHEAL on 100 mm visual analogue scales. Total scores range from 0 -100. Higher scores reflect higher levels of confidence.
Changes in Coercive Control on the Women's Experiences of Battering Scale (WEB) | Baseline, 6 months
  10 item self-report measure of the intensity of coercive control experienced by women in response to intimate partner violence. Total scores range from 10 to 60. Higher scores reflect higher levels of experiences of coercive control.
Changes in Coercive Control on the Women's Experiences of Battering Scale (WEB) | Baseline, 12 months
  10 item self-report measure of the intensity of coercive control experienced by women in response to intimate partner violence. Total scores range from 10 to 60. Higher scores reflect higher levels of experiences of coercive control.
Changes in Coercive Control on the Women's Experiences of Battering Scale (WEB) | Baseline, 18 months
  10 item self-report measure of the intensity of coercive control experienced by women in response to intimate partner violence. Total scores range from 10-60. Higher scores reflect higher levels of experiences of coercive control.

OTHER OUTCOMES:
Severity of Intimate Partner Violence on the Composite Abuse Scale Revised - Short Form (CASr-SF) | Baseline, 6, 12, 18 months
  15 item validated measure of severity of intimate partner violence
Problem Drinking on the AUDIT | Baseline, 6, 12, 18 months
  Self-report measure of alcohol mis-use

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn Ford-Gilboe, PhD, Principal Investigator — Western University
Locations (3):
- Canada (3):
  - University of British Columbia, Vancouver, British Columbia
  - University of New Brunswick, Fredericton, New Brunswick
  - Western University, London, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ford-Gilboe M, Varcoe C, Scott-Storey K, Browne AJ, Jack SM, Jackson K, Mantler T, O'Donnell S, Patten-Lu N, Smye V, Wathen CN, Perrin N. Longitudinal effectiveness of a woman-led, nurse delivered health promotion intervention for women who have experienced intimate partner violence: iHEAL randomized controlled trial. BMC Public Health. 2024 Feb 7;24(1):398. doi: 10.1186/s12889-023-17578-4. PMID 38326832